CLINICAL TRIAL: NCT00587990
Title: A Phase I/II, Randomized, Double-Blinded, Placebo-Controlled Study of the Safety and Efficacy of Intramyocardial Injection of Autologous Human Mesenchymal Stem Cells (MSCs) in Patients With Chronic Ischemic Left Ventricular Dysfunction Secondary to Myocardial Infarction (MI) Undergoing Cardiac Surgery for Coronary Artery Bypass Grafting (CABG)
Brief Title: Prospective Randomized Study of Mesenchymal Stem Cell Therapy in Patients Undergoing Cardiac Surgery (PROMETHEUS)
Acronym: PROMETHEUS
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Difficulty in recruitment.
Sponsor: Joshua M Hare (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Johns Hopkins University Specialized Center for Cell Based Therapy (Other); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor-Investigator, Joshua M Hare, Director, Interdisciplinary Stem Cell Institute, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20070598; U54HL081028 (NIH)
Record Dates: First submitted 2008-01-02; First posted 2008-01-08 (Estimated); Results first posted 2015-04-02 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Stem Cell Transplantation; Ventricular Dysfunction, Left
Keywords: Chronic Ischemic Left Ventricular Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Left | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lower dose mesenchymal stem cell (MSC) injection (Experimental): Participants will receive lower dose mesenchymal stem cell injections for a total of 2 x 10^7 cells
  Interventions: Biological: Lower dose mesenchymal stem cell (MSC) injection
- Higher dose MSC injection (Experimental): Participants will receive higher dose of mesenchymal stem cell injections for a total of 2 x 10^8 cells
  Interventions: Biological: Higher dose MSC injection
- (3) Placebo (Placebo Comparator): Participants will receive placebo injections
  Interventions: Genetic: Placebo

INTERVENTIONS:
Biological: Lower dose mesenchymal stem cell (MSC) injection — Participants will receive between 10 and 20 intramyocardial injections of 2 million MSCs per 0.25-0.5 cubic centimeter (cc) for a total of 2 x 10^7 cells. The injections will be administered following completion of CABG surgery.
  Arms: Lower dose mesenchymal stem cell (MSC) injection
Genetic: Placebo — Participants will receive between 10 and 20 placebo injections that consist of phosphate buffered saline (PBS) and 1% human serum albumin (HSA).
  Arms: (3) Placebo
Biological: Higher dose MSC injection — Participants will receive between 10 and 20 intramyocardial injections of 20 million MSCs per 0.25-0.5 cc for a total of 2 x 10^8 cells. The injections will be administered following completion of CABG surgery.
  Arms: Higher dose MSC injection

SUMMARY:
Heart attacks are a leading cause of death in both men and women in the United States. When a person has a heart attack, blood is unable to reach a certain area of the heart, and if the blood supply is not re-established quickly, that area of the heart can suffer permanent damage. While recovery from a heart attack can be managed through medications and lifestyle changes, these treatments can not reverse the original damage to the heart. Current research is focusing on the development of cell-based therapies using stem cells to repair organs that have been irreversibly damaged by disease. A specific form of stem cells, called adult mesenchymal stem cells (MSCs), has shown promise for heart repair. This study will evaluate the safety and effectiveness of injecting MSCs into the heart to repair and restore heart function in people who have had a heart attack and who are having heart surgery for coronary artery bypass grafting (CABG).

DETAILED DESCRIPTION:
Participation in this study will last 18 months. Potential participants will undergo initial screening 5 to 7 weeks prior to CABG surgery. Screening will include a physical exam, blood draw, pregnancy test, questions about medical history, current medications, and alcohol or drug use, an electrocardiogram (ECG), magnetic resonance imaging (MRI) of the heart, questionnaires, an echocardiogram and a computed tomography (CT) scan. Eligible participants will then undergo two baseline visits within 6 weeks of their scheduled surgery. Baseline Visit 1 will consist of vital sign measurements, a bone marrow aspiration to obtain MSCs and a blood draw for a biomarker test. Baseline Visit 2 will include treadmill test, 6-minute walk test, pulmonary function (FEV1) study and a 48 Hour Ambulatory ECG. After the second baseline visit, participants will be assigned randomly to receive either MSCs or placebo after surgery.

On the day of surgery, once all of the bypass grafts have been placed, a high or low dose of MSCs or placebo will be injected into a damaged area of the heart that did not receive a bypass graft. After receiving the injections, participants will remain in the hospital for up to 7 days. During this stay, participants will undergo a daily blood draw, urine test, ECG, and ambulatory ECG monitoring for the first 96 hours after surgery.

Upon being discharged, participants will return for monthly visits for 6 months and for follow-up visits 12 and 18 months after surgery. These visits will repeat most initial screening and baseline tests. There will be one additional visit 14 days after surgery, which will include questions about side effects, a physical exam, and a 48-hour ambulatory ECG.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic ischemic heart failure caused by a heart attack
* Scheduled to undergo cardiac surgery for CABG
* Ejection fraction between 15% and 50%
* Presence of an akinetic or dyskinetic region by standard imaging

Exclusion Criteria:

* Glomerular filtration rate of less than 50 mL/min/1.73m2 at study entry
* Contraindication to performance of an MRI scan
* Bone marrow dysfunction, as evidenced by a 20% or more deviation from normal hematocrit, white blood cell count, or platelet values without another explanation
* A coagulopathy condition not due to a reversible cause (i.e., Coumadin)
* Known, serious radiographic contrast allergy
* Known allergies to penicillin or streptomycin
* Organ transplant recipient
* Clinical history of malignancy within 5 years of study entry (e.g., patients with prior malignancy must be disease free for 5 years), except curatively treated basal cell carcinoma, squamous cell carcinoma, or cervical carcinoma
* Non-cardiac condition that limits lifespan to less than 1 year
* On chronic therapy with immunosuppressant medication
* Serum positive for HIV, hepatitis B, or hepatitis C
* Female who is pregnant, nursing, or of child-bearing potential and not practicing effective birth control methods

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua M. Hare, MD, Principal Investigator — University of Miami; Gary Gerstenblith, MD, Principal Investigator — Johns Hopkins University; John V. Conte, MD, Principal Investigator — Johns Hopkins University; Steven P. Schulman, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - University of Miami Miller School of Medicine, Miami, Florida
  - Johns Hopkins University School of Medicine, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Karantalis V, DiFede DL, Gerstenblith G, Pham S, Symes J, Zambrano JP, Fishman J, Pattany P, McNiece I, Conte J, Schulman S, Wu K, Shah A, Breton E, Davis-Sproul J, Schwarz R, Feigenbaum G, Mushtaq M, Suncion VY, Lardo AC, Borrello I, Mendizabal A, Karas TZ, Byrnes J, Lowery M, Heldman AW, Hare JM. Autologous mesenchymal stem cells produce concordant improvements in regional function, tissue perfusion, and fibrotic burden when administered to patients undergoing coronary artery bypass grafting: The Prospective Randomized Study of Mesenchymal Stem Cell Therapy in Patients Undergoing Cardiac Surgery (PROMETHEUS) trial. Circ Res. 2014 Apr 11;114(8):1302-10. doi: 10.1161/CIRCRESAHA.114.303180. Epub 2014 Feb 24. PMID 24565698

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This trial, which originally was designed to enroll 45 patients, was suspended after 9 patients were enrolled because of slow accrual.
Groups:
- (1) Lower MSC Dose: Participants will receive lower dose mesenchymal stem cell injections for a total of 2 x 107 cells
  Lower dose mesenchymal stem cell (MSC) injection: Participants will receive between 10 and 20 intramyocardial injections of 2 million MSCs per 0.25-0.5 cubic centimeter (cc) for a total of 2 x 107 cells. The injections will be administered following completion of CABG surgery.
- (2) Higher MSC Dose: Participants will receive higher dose of mesenchymal stem cell injections for a total of 2 x 108 cells
  Higher dose MSC injection: Participants will receive between 10 and 20 intramyocardial injections of 20 million MSCs per 0.25-0.5 cc for a total of 2 x 108 cells. The injections will be administered following completion of CABG surgery.
- (3) Placebo Injection: Participants will receive placebo injections
  Placebo: Participants will receive between 10 and 20 placebo injections that consist of phosphate buffered saline (PBS) and 1% human serum albumin (HSA).
Period: Overall Study
Arm/Group | (1) Lower MSC Dose | (2) Higher MSC Dose | (3) Placebo Injection
Started | 2 | 4 | 3
Completed | 2 | 4 | 2
Not Completed | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | (1) Lower MSC Dose | (2) Higher MSC Dose | (3) Placebo | Total
Number analyzed (Participants) | 2 | 4 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3668720 (13.4742319) | 51.9240246 (9.1760352) | 63.6276523 (2.9733072) | 57.7014222 (9.3869460)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 2 | 4 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Serious Adverse Events
Description: Six-month post-CABG surgery serious adverse event (SAE) proportion of patients experiencing a composite of sustained ventricular arrhythmias, (lasting longer than 15 seconds), with hemodynamic compromise, sudden unexpected death at six months, ectopic tissue formation at 12 months by chest/abdomen/pelvis CT exam.
Time Frame: 12 Months
Population: Due to the early termination of the study, there was an insufficient sample size of the Low and High dose of MSCs participants. The statistical analysis plan was revised to combine the low and high dose groups in order to make a comparison to the participants who received a placebo.
Measure: Count of Participants; unit: Participants
Groups:
- Treated Group (Low/High Doses): Participants who received mesenchymal stem cell injections.
- Placebo Group: Participants who received placebo injections.
Arm/Group | Treated Group (Low/High Doses) | Placebo Group
Number analyzed (Participants) | 6 | 3
Participants | 0 | 1

2. Secondary Outcome: Change in Infarct Scar Size (ISS) Over 18 Month Period
Description: Change in infarct scar size (ISS) between baseline and 6-month and 18 month visits as determined by delayed contrast-enhanced MRI.
Time Frame: Baseline, 6 Months, 18 Months
Population: One placebo subject expired Day 3 post injection. Due to the early termination of the study, there was an insufficient sample size of the Low and High dose of MSCs participants. The statistical analysis plan was revised to combine the low and high dose groups in order to make a comparison to the participants who received a placebo.
Measure: Mean (95% Confidence Interval); unit: Grams (g)
Arm/Group | Treated Group (Low/High Doses) | Placebo Group
Number analyzed (Participants) | 6 | 2
Grams (g)
  6 Months | -2.37 [-5.64 to .89] | -2.16 [-40.53 to 36.21]
  18 Months: number analyzed (Participants) | 5 | 2
  18 Months | -5.91 [-8.85 to -2.97] | -5.32 [-78.25 to 67.61]

3. Secondary Outcome: Left Ventricular Function (LVF) in Region of MSC Injection
Description: The Left Ventricular Function differences in the region of MSC injection were evaluated. LVF is evaluated via ECHO as the percentage of ejected blood.
Time Frame: Assessed at Baseline and 18 Months
Population: Due to the early termination of the study, there was an insufficient sample size of the Low and High dose of MSCs participants. The statistical analysis plan was revised to combine the low and high dose groups in order to make a comparison to the participants who received a placebo. One placebo subject expired Day 3 post injection.
Measure: Mean (Standard Error); unit: percentage of ejected blood
Arm/Group | Treated Group (Low/High Doses) | Placebo Group
Number analyzed (Participants) | 6 | 2
percentage of ejected blood
  Baseline | -15.26 (3.15) | -18.53 (2.71)
  18 Months | -21.13 (1.68) | -19.66 (1.07)

4. Secondary Outcome: Regional Left Ventricular Wall Thickening
Description: Difference between baseline and 18 month regional left ventricular wall thickening as determined by MRI.
Time Frame: Assessed at Baseline and 18 months
Population: Due to the early termination of the study, there was an insufficient sample size of the Low and High dose of MSCs participants. The statistical analysis plan was revised to combine the low and high dose groups in order to make a comparison to the participants who received a placebo.One placebo subject expired Day 3 post injection.
Measure: Mean (Standard Error); unit: mm
Arm/Group | Treated Group (Low/High Doses) | Placebo Group
Number analyzed (Participants) | 6 | 2
mm
  Baseline | 20.68 (6.67) | 32.21 (9.97)
  18 Months | 47.87 (9.45) | 42.09 (9.49)

5. Secondary Outcome: Left Ventricular End Diastolic Wall Thickness
Description: Difference between the baseline and 18 month left ventricular end diastolic wall thickness as determined by MRI and echocardiogram.
Time Frame: Assessed at Baseline and 18 months
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mm
Arm/Group | Treated Group (Low/High Doses) | Placebo Group
Number analyzed (Participants) | 6 | 2
mm
  Baseline | 5.86 (.46) | 16.15 (2.72)
  18 Months | 6.17 (.48) | 18.54 (1.55)

6. Secondary Outcome: Change in Left Ventricular End Diastolic and Systolic Volume
Description: Change in left ventricular end diastolic and systolic volume as determined by MRI and echocardiogram.
Time Frame: Baseline, 6 Months, 18 Months
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: ml
Arm/Group | Treated Group (Low/High Doses) | Placebo Group
Number analyzed (Participants) | 6 | 2
ml
  End Diastolic Volume from Baseline to 6 Months | 192.92 [115.91 to 281.93] | 169.63 [-468.29 to 807.54]
  End Diastolic from 6 Month to 18 Month | 218.73 [98.85 to 338.61] | 172.01 [-245.46 to 589.47]
  End Systolic Volume from Baseline to 6 Months | 130.09 [46.47 to 213.71] | 97.13 [-416.33 to 610.59]
  End Systolic from 6 Month to 18 Month | 135.99 [29.07 to 242.90] | 94.90 [-307.45 to 497.24]

7. Secondary Outcome: Change in Left Ventricular Ejection Fraction
Description: Change between baseline to 6-month and 18-month left ventricular ejection fraction (LVEF) as determined by MRI and echocardiogram.
Time Frame: Baseline to 6 Months, Baseline to 18 Months
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: percentage of Ejection Fraction
Arm/Group | Treated Group (Low/High Doses) | Placebo Group
Number analyzed (Participants) | 6 | 2
percentage of Ejection Fraction
  Baseline to 6 Months | -.34 [-6.6 to 5.92] | 13.18 [-68.65 to 95.01]
  Baseline to 18 Months | 2.50 [-3.35 to 8.34] | 14.61 [-59.15 to 88.36]

8. Secondary Outcome: Change in Peak Volume Oxygen
Description: Change in Peak VO2 as determined by treadmill test (mL/mg/min) from Baseline to 6 and from baseline to 18 months
Time Frame: Baseline, 6 Months, 18 Months
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: (mL/mg/min)
Arm/Group | Treated Group (Low/High Doses) | Placebo Group
Number analyzed (Participants) | 6 | 2
(mL/mg/min)
  Baseline to 6 Months | .2 [-1.1 to 1.4] | -.2 [-12.9 to 12.5]
  Baseline to 18 Months | -.2 [-1.8 to 1.3] | -.4 [-10.6 to 9.8]

9. Secondary Outcome: Change in Six Minute Walk Test
Description: Change in Six Minute Walk Test (in meters) from Baseline to 6 Months and Baseline to 18 Months
Time Frame: Baseline, 6 Months, 18 Months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Meters
Arm/Group | Treated Group (Low/High Doses) | Placebo Group
Number analyzed (Participants) | 6 | 2
Meters
  Baseline to 6 Months | 67 [-453.0 to 309.0] | -30.00 [-30.00 to -30.00]
  Baseline to 18 Months | 67 [-199.0 to 309.0] | -33.0 [-36 to -30]

10. Secondary Outcome: Change in NYHA Functional Class
Description: Change in New York Heart Association (NYHA) Functional Classification based on patient's self reported activity level.
  Worsened: documented increase in limitations of physical activity as self-described by subject Improved: documented decrease in limitations of physical activity as self-described by subject Unchanged: no documented change in limitations of physical activity as self-described by subject
Time Frame: Baseline to 6 Months, 6 months to 18 Months
Population: Due to the early termination of the study,there was an insufficient sample size of the MSC treated participants.The statistical analysis plan was revised to combine the low and high dose groups.1 treated subject's NYHA class was not captured at the 18 Month time point.1 placebo treated subject expired prior to 6 and 18 months NYHA class assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Group (Low/High Doses) | Placebo Group
Number analyzed (Participants) | 6 | 3
Participants
  Baseline to 6 Months, Worsened: number analyzed (Participants) | 6 | 2
  Baseline to 6 Months, Worsened | 0 | 0
  Baseline to 6 Months, Improved: number analyzed (Participants) | 6 | 2
  Baseline to 6 Months, Improved | 3 | 1
  Baseline to 6 Months, Unchanged: number analyzed (Participants) | 6 | 2
  Baseline to 6 Months, Unchanged | 3 | 1
  6 Months to 18 Months, Worsened: number analyzed (Participants) | 5 | 2
  6 Months to 18 Months, Worsened | 2 | 0
  6 Months to 18 Months, Improved: number analyzed (Participants) | 5 | 2
  6 Months to 18 Months, Improved | 0 | 1
  6 Months to 18 Months, Unchanged: number analyzed (Participants) | 5 | 2
  6 Months to 18 Months, Unchanged | 3 | 1

11. Secondary Outcome: Minnesota Living With Heart Failure Questionnaire Scores
Description: Minnesota Living with Heart Failure (MLHF) questionnaire has a total score from 0 to 105. A higher score indicates that participants heart failure is preventing them from living their lives measured at two time points.
Time Frame: Assessed at 6 Months and 18 Months
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Treated Group (Low/High Doses) | Placebo Group
Number analyzed (Participants) | 6 | 2
score on a scale
  6 Month Visit | 11.5 [-10.8 to 33.8] | 54.5 [-66.2 to 175.2]
  18 Month Visit | 7.3 [-3.6 to 18.3] | 10.5 [-122.9 to 143.9]

12. Secondary Outcome: Incidence of Major Adverse Cardiac Events (MACE)
Description: Incidence of Major Adverse Cardiac Events (MACE). A composite incidence of (1) death, (2) hospitalization for heart failure, or (3) non-fatal recurrent Ml.
Time Frame: 18 Months
Population: as for outcome 1
Measure: Number; unit: # of Major Adverse Cardiac Events (MACE)
Arm/Group | Treated Group (Low/High Doses) | Placebo Group
Number analyzed (Participants) | 6 | 3
# of Major Adverse Cardiac Events (MACE) | 0 | 1

13. Secondary Outcome: Number of Participants With Abnormal 48-Hour Ambulatory ECG Recordings
Description: Ambulatory ECG monitoring is the most widely employed technology for the evaluation of a patient with symptoms suggestive of cardiac arrhythmia or conduction abnormality.
  When the patient returns for follow up the 48- Hour Ambulatory monitor provides the data to the site staff to detect any abnormal recordings based upon standard ECG protocol.
Time Frame: Assessed at 6 Months, 12 Months, and 18 Months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Treated Group (Low/High Doses) | Placebo Group
Number analyzed (Participants) | 6 | 2
Participants
  6 Month Visit | 4 | 2
  12 Month Visit: number analyzed (Participants) | 3 | 2
  12 Month Visit | 3 | 2
  18 Month Visit: number analyzed (Participants) | 5 | 2
  18 Month Visit | 5 | 2

14. Secondary Outcome: Change in Pulmonary Function
Description: Change in Pulmonary Function from Baseline to 6 month, Baseline to 12 month, and Baseline to 18 month visits as measured by forced expiratory volume in 1 second (FEV1)
Time Frame: Baseline, 6 Months, 12 Months, 18 Months
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | Treated Group (Low/High Doses) | Placebo Group
Number analyzed (Participants) | 6 | 2
Liters
  Baseline to 6 Months | -7.2 [-16.3 to 1.9] | 7.0 [-81.9 to 95.9]
  Baseline to 12 Months | -8.5 [-18.9 to 1.9] | -5.5 [-62.7 to 51.7]
  Baseline to 18 Months | -7.2 [-23.1 to 8.8] | 7.5 [-176.7 to 191.7]

15. Secondary Outcome: Serial Troponin Values (ng/mL)
Description: Serial Troponin Values (ng/mL) Values from Baseline to 48 Hours Post CABG
Time Frame: Assessed at Baseline, 12 hours, 24 hours, 36 hours, and 48 hours post CABG
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: ng/mL
Arm/Group | Treated Group (Low/High Doses) | Placebo Group
Number analyzed (Participants) | 6 | 3
ng/mL
  Baseline | .01 [.01 to .25] | .01 [0 to .01]
  12H | .76 [.03 to 2.0] | .76 [.18 to 1.26]
  24H | .35 [.16 to 3.31] | .1 [.03 to .49]
  36H | .55 [.23 to 2.23] | .36 [.13 to 1.57]
  48H | .21 [.14 to 4.44] | .2 [.2 to .2]

16. Secondary Outcome: Creatinine Kinase - Muscle/Brain (MB) (ng/mL)
Description: Creatinine Kinase MB (ng/mL) Values every 12 hours from Baseline to 48 Hours Post CABG
Time Frame: Assessed at Baseline, 12 Hours, 24 Hours, 36 Hours, and 48 hours post CABG
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: ng/mL
Arm/Group | Treated Group (Low/High Doses) | Placebo Group
Number analyzed (Participants) | 6 | 3
ng/mL
  Baseline | 2.2 [.7 to 8.10] | 2.6 [2.44 to 3.00]
  12H | 19.6 [9 to 32.10] | 24.75 [16.9 to 30.8]
  24H | 12.39 [3 to 21.60] | 15.5 [11.5 to 66.28]
  36H | 8.04 [1 to 11.80] | 8.1 [7.5 to 99.99]
  48H | 4.75 [2 to 8.99] | 6 [6 to 6]

17. Secondary Outcome: Number of Clinically Significant Laboratory Values
Description: Clinically significant laboratory values are first determined via standard laboratory normal values from a CAP and CLIA certified Laboratory and then assessed by investigator based on specific patient conditions and disease state.
Time Frame: 18 Months
Population: as for outcome 3
Measure: Number; unit: Incidents
Arm/Group | Treated Group (Low/High Doses) | Placebo Group
Number analyzed (Participants) | 6 | 2
Incidents
  Clinically Significant Hematology Values | 6 | 0
  Clinically Significant Clinical Chemistry Values | 9 | 0
  Clinically Significant Urinalysis Values | 0 | 0

18. Secondary Outcome: Rate of Treatment Emergent Adverse Events
Description: Rate of Treatment Emergent Adverse Events Post Coronary Artery Bypass Graft (CABG) at 6 Months, 12 Months, and 18 Months
Time Frame: Assessed at 6 Months, 12 Months, and 18 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Number of Adverse Events
Arm/Group | Treated Group (Low/High Doses) | Placebo Group
Number analyzed (Participants) | 6 | 3
Number of Adverse Events
  6 Months Post CABG | 9.5 [1 to 30] | 5.0 [1 to 10]
  12 Months Post CABG | 10.0 [1 to 33] | 5.7 [1 to 11]
  18 Months Post CABG | 11 [1 to 36] | 6 [1 to 11]

19. Secondary Outcome: Number of Abnormal Echocardiogram Readings 2 Days Post CABG.
Description: The number of abnormal Echocardiogram readings 2 Days Post CABG will be documented based on transthoracic Echocardiographic standards. However, although Echocardiograms 2 days post CABG operation may show abnormalities which is standard in this population, this testing is instrumental because it measures End- diastolic wall thickness and Left ventricular volumes at end-diastole and end-systole.
Time Frame: Day 2
Population: Due to the early termination of the study, there was an insufficient sample size of the Low and High dose of MSCs participants. The statistical analysis plan was revised to combine dose groups to make a comparison to placebo subjects.
Measure: Number; unit: Abnormal Echocardiograms
Arm/Group | Treated Group (Low/High Doses) | Placebo Group
Number analyzed (Participants) | 6 | 3
Abnormal Echocardiograms | 6 | 3

ADVERSE EVENTS:
Time Frame: 18 Months
Arm/Group | (1) Lower MSC Dose | (2) Higher MSC Dose | (3) Placebo Injection
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4 | 1/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 2/4 | 3/3
Other Adverse Events (participants affected / at risk) | 2/2 | 4/4 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | (1) Lower MSC Dose (N=2) | (2) Higher MSC Dose (N=4) | (3) Placebo Injection (N=3)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (3)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural site reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Debridement (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Ischemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | (1) Lower MSC Dose (N=2) | (2) Higher MSC Dose (N=4) | (3) Placebo Injection (N=3)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Tenderness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Back Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood triglycerides abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hematocrit decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (3) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Ageusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Erection increased (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hematoma evacuation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations due to slow enrollment and premature closure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes